CLINICAL TRIAL: NCT03987698
Title: Phase II Clinical Study of PD-1 Monoclonal Antibody Combination With Autologous Cytokine-induced Killer Cell Immunotherapy in the Second-line Treatment of Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Study of PD-1 Inhibitor Combination With Autologous Cell Immunotherapy in the Metastatic Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2017232
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — camrelizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: CIK+PD-1i (Experimental): SHR-1210 & CIK cells
  SHR-1210,200mg/d,intravenous infusion,d1; CIK cells, 1x10^10 (10 billion ), intravenous infusion,d14; Q3W.
  Interventions: Biological: SHR-1210; Biological: CIK cells
- Arm 2: Control (Active Comparator): SHR-1210,200mg/d,intravenous infusion,d1; Q3W.
  Interventions: Biological: SHR-1210

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 injection
  Other Names: PD-1 inhibitor
Biological: CIK cells — CIK cells injection
  Other Names: Cytokine-induced killer cells
  Arms: Arm 1: CIK+PD-1i

SUMMARY:
This randomized, multicenter,open-label, phase II study is to evaluate the effects of PD-1 inhibitor combination with autologous cytokine-induced killer cell immunotherapy in the second-line treatment of patients with metastatic clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
In the experimental group, patients received Camrelizumab injection (SHR-1210) 200mg d1, CIK cells 1x10^10 d14; Q3W, for 4 cycles; then Camrelizumab injection maintenance treatment for 2 years. In the control group, patients received Camrelizumab injection 200mg d1, Q3W, for 2 years.

ELIGIBILITY:
Inclusion Criteria:

Subjects who must meet all the following criteria should be selected:

1. Agreeing to participate in this study and signing a written informed consent.
2. Male or female,from 18 to 75 years (including 18 and 75 years).
3. The life expectancy will be longer than 3 months and can be followed up.
4. Patients with metastatic clear cell renal cell carcinoma were confirmed by histological /cytological and imaging examinations. According to RECIST 1.1 standard, there will be at least one measurable lesion.
5. Patients with disease progression after treatment with interferon or TKI.
6. ECOG score will be 0 or 1 within 7 days before randomization.
7. Within 14 days before the start of treatment, the results of laboratory test of blood routine, liver, kidney function and hormone levels must be met the following criteria:

   White blood cells: more than 3.0 × 109/L; Platelets: more than 100 × 109/L; Neutrophils: more than 1.5 × 109/L; Hemoglobin: more than 80g/L; Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN); Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN; Serum bilirubin: less than 1.25 × ULN; Serum creatinine: less than 1.25 × ULN. Cortisol and thyroid function will be in the normal range.
8. The toxicity and side effects of previous chemotherapy will must be alleviated to grade 1 or below (except hair loss).
9. Female subjects must take effective contraceptive measures throughout the study period; serum or urine pregnancy test results must be negative during screening and the whole study period.
10. Male subjects should take effective contraceptive measures from the beginning of treatment to within 6 months after the end of treatment.

Exclusion Criteria:

Subjects who meet any of the following criteria could not participate in this study:

1. Other malignant tumors needed treatment within five years.
2. Allogeneic tissue/organ transplantation.
3. Participating in research drug therapy within 4 weeks before the first administration of the trial.
4. Systemic glucocorticoid therapy or any other form of immunosuppressive therapy (except glucocorticoid preconditioned with docetaxel) is being administered within 3 days before the first administration of the experimental therapy.
5. Received anti-tumor monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy or major surgery within 4 weeks before the first use of the drug; received chest radiotherapy greater than 30 Gy within 6 months before the first use of the drug; and received chest radiotherapy with 30 Gy or less within 1 month before the first use of the drug.
6. Previous treatment with PD-1/PD-L1 antibodies.
7. Over the past two years, patients with active autoimmune diseases requiring systemic treatment, such as the use of corticosteroids, or immunosuppressants. Substitution therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction) is not a systemic treatment.
8. Patients with congenital or acquired immunodeficiency (e.g. HIV-infected persons), active hepatitis B (HBV-DNA > 10^3 copies/ml) or hepatitis C (hepatitis C antibody positive), and HCV-RNA higher than the detection limit of the analytical method.
9. Subjects with active central nervous system (CNS) metastases and/or cancerous meningitis.
10. Patients with active infections requiring systemic intravenous therapy.
11. Mental illness or other illnesses, such as uncontrollable heart disease or pulmonary disease, diabetes, etc.
12. Subjects who are known to be allergic to any of the constituents of the drug being studied.
13. Subjects with a recent history of drug abuse (including alcohol) within one year.
14. Compliance is poor and can not cooperate with clinical research.
15. Female subjects who are pregnant or breastfeeding, or who are expected to be pregnant during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 year
  PFS will be calculated from initiation of treatment until first progression, and patients alive in stable state will be censored at the time of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Xiubao Ren, MD. PhD., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Li S, Qin J, Sun Q, Zhao H, Xiong Y, Wang Y, Han Y, Zhang J, Zhang W, Shen M, Yang F, Ren B, Zhou L, Li R, Hui Z, Tian X, Cao S, Du W, Yu W, Liu L, Zhang X, Ren X. Randomized pilot study of camrelizumab with or without autologous cytokine-induced killer cells in refractory clear cell renal cell carcinoma. Sci Rep. 2026 Feb 7. doi: 10.1038/s41598-026-38881-1. Online ahead of print. PMID 41654611